CLINICAL TRIAL: NCT02993588
Title: Impact of Melatonin Adjuvant Therapy on IVF/ICSI Outcomes in Prospective Poor Responders: A Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Impact of Melatonin on IVF/ICSI Outcomes in Prospective Poor Responders
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Saber Thabet Abdalmageed, Lecturer of OBGYN, Women Health Hospital, Assiut Univerisity, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Melatonin RCT
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: In Vitro Fertilization; Poor Ovarian Response
Keywords: Melatonin; IVF/ICSI; Poor ovarian response
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melatonin (Experimental): Melatonin 6 mg tablet once daily.
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo tablet once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin 6 mg tablet once daily
  Arms: Melatonin
Other: Placebo — one tablet once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the impact of melatonin administration on in vitro fertilization (IVF/ICSI) outcomes namely the total number and quality of the oocytes and embryos in the prospective poor responders.

DETAILED DESCRIPTION:
The prospective poor responders have been associated with lower number and poorer oocyte quality. Melatonin is suggested to have antioxidative effects which may contribute to improving the IVF/ICSI outcomes in this group of patients who expected to have poor outcomes. However, the expected beneficial effects of melatonin have not yet been investigated. The purpose of this study is to investigate the impact of melatonin administration on IVF/ICSI outcomes namely the total number and quality of the oocytes and embryos in the prospective poor responders. A randomized, double-blinded, placebo-controlled study is used to investigate the impact of melatonin on the IVF/ICSI outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Prospective poor responder with AMH < 1 ng/ml and AFC < 8 (in both ovaries).

Exclusion Criteria:

* Severe male factor infertility.

Ages: 30 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Total number of retrieved mature oocytes | On the day of oocyte retrieval procedure

CONTACTS AND LOCATIONS:
Overall Officials: Osama Abdalmageed, MD, Principal Investigator — Women health center
Locations (2):
- Egypt (2):
  - Osama Abdalmageed, Asyut, Asyut Governorate
  - Osama Abdalmageed, Asyut, Non-US/Non-Canadian

IPD SHARING:
Plan to Share IPD: No
The data will be kept with the study team only and it is not allowed by our institution regulations to share the data.

REFERENCES:
- [Background] Fernando S, Rombauts L. Melatonin: shedding light on infertility?--A review of the recent literature. J Ovarian Res. 2014 Oct 21;7:98. doi: 10.1186/s13048-014-0098-y. PMID 25330986